CLINICAL TRIAL: NCT06382168
Title: Phase I/II Study of DFP-10917 in Combination With Venetoclax in Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: DFP-10917 in Combination With Venetoclax in Relapsed or Refractory Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Delta-Fly Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D19-11186
Expanded Access: Available
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2024-09

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — DFP-10917; venetoclax

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DFP-10917 + Venetoclax for 14 days (Experimental): DFP-10917 4 mg/m^2/day with venetoclax 400 mg once daily for 14 days
  Interventions: Drug: DFP-10917; Drug: Venetoclax
- DFP-10917 + Venetoclax for 10 days (Experimental): DFP-10917 4 mg/m^2/day with venetoclax 400 mg once daily for 10 days
  Interventions: Drug: DFP-10917; Drug: Venetoclax

INTERVENTIONS:
Drug: DFP-10917 — DFP-10917 4 mg/m^2/day is given as a continuous 14-day intravenous infusion, followed by a 14-day rest in each 28-day cycle.
Drug: Venetoclax — Venetoclax 400 mg once daily for 10-14 days, followed by a 14-day rest in each 28-day cycle.

SUMMARY:
This Phase I/II trial evaluates the safety and preliminary efficacy of DFP-10917 combined with venetoclax in relapsed or refractory acute myeloid leukemia. DFP-10917 is given as a 14-day continuous IV infusion every 28 days, alongside a 14-day oral course of venetoclax following an initial dose ramp-up. The initial phase tests a starting dose of 4 mg/m²/day of DFP-10917 with 400 mg daily of venetoclax. The Data Monitoring Committee reviews toxicity after one treatment cycle. If DLTs are minimal, more patients are added to confirm safety. If the lower dose level shows tolerability, it proceeds to the Phase II expansion to assess the treatment's effectiveness against leukemia using a Simon's two-stage design, targeting up to 17 participants.

DETAILED DESCRIPTION:
This study is a Phase I/II, open-label trial exploring dosage and expansion cohorts to assess the safety and preliminary efficacy of DFP-10917 in combination with venetoclax for patients with relapsed or refractory acute myeloid leukemia (AML). DFP-10917 will be administered as a 14-day continuous intravenous infusion starting on Day 1, followed by a 14-day rest period, during each 28-day cycle. This will occur concurrently with venetoclax, administered orally at a dose of 400 mg daily for 14 days following a dose ramp-up phase (100 mg and 200 mg on Day 1 and 2, respectively).

In Phase I, the starting dose for DFP-10917 is 4 mg/m²/day, administered concurrently with 400 mg of venetoclax once daily for 14 days (Dose Level 1). The Data Monitoring Committee (DMC) will assess dose-limiting toxicities (DLTs) after three patients are enrolled at this dose level and the last patient has completed the 4-week safety assessment period (i.e., one cycle of the combination regimen). At Dose Level 1 (4 mg/m²/day of DFP-10917 with venetoclax 400 mg daily for 14 days), if none of the three patients experience a DLT, the study will enroll an additional three patients at this dose level to confirm the combination's safety and tolerability. If one out of three patients experiences a DLT, up to three additional patients may be enrolled. If one or fewer out of six treated patients experience a DLT at Dose Level 1, this dose will be declared the recommended Phase II dose (RP2D) and used in the Phase II expansion cohort. If two or more patients out of the total three to six patients at Dose Level 1 experience a DLT, the study will continue enrollment at Dose Level 1 (4 mg/m²/day of DFP-10917 for 14 days concurrently with venetoclax 400 mg daily for 10 days of each 28-day cycle) to determine the safety and tolerability of Dose Level -1. A patient who discontinues therapy during Cycle 1 without experiencing DLTs is considered evaluable for safety purposes only if all scheduled doses of DFP-10917 and at least 80% of the venetoclax doses were administered in the first cycle. Once the RP2D of DFP-10917 in combination with venetoclax is determined, the expansion cohort will begin enrollment to evaluate the anti-leukemia efficacy of this combination. A Simon's two-stage min-max design will be employed, with up to 17 patients expected to participate.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent and ability to comply with protocol requirements.
* Histologically or pathologically confirmed diagnosis of acute myeloid leukemia based on World Health Organization classification that has relapsed after, or is refractory to, up to 2 prior induction regimens that may have included intensive chemotherapy (e.g., "7+3" cytarabine and daunorubicin), epigenetic therapy (i.e., azacitidine or decitabine with/without venetoclax), or targeted therapy (e.g., FLT-3, IDH 1/2, BCL-2, monoclonal antibody).

(Relapse is defined as reemergence of ≥5% leukemia blasts in bone marrow or ≥1% blasts in peripheral blood 90 days to 24 months after first complete remission or complete remission with incomplete hematologic recovery. Refractory acute myeloid leukemia is defined as persistent disease ≥28 days after initiation of intensive induction therapy (up to 2 induction cycles) or relapse <90 days after first complete remission or complete remission with incomplete hematologic recover. Refractory disease for patients undergoing hypomethylating agent induction is defined as lack of remission following at least 2 cycles of epigenetic therapy without reduction in bone marrow blast status).

* Adequate organ function as defined by the following laboratory values:

  * Creatinine clearance >30 mL/min (by Cockcroft-Gault method),
  * Total serum bilirubin <1.5 × upper limit of normal unless due to Gilbert's syndrome, leukemic organ involvement, hemolysis or considered an effect of regular blood transfusions,
  * Alanine aminotransferase and aspartate aminotransferase <3 × upper limit of normal, unless due to leukemic organ involvement.
* Eastern Cooperative Oncology Group performance status of 0, 1, or 2).
* Projected life expectancy of ≥12 weeks.
* Female patients of childbearing potential must:

  * Have a negative serum or urine pregnancy test prior to study treatment initiation.
  * Agree to use at least 1 highly effective form of contraception during study treatment and for 3 months after the last dose.
* Male patients with female partners of childbearing potential must -- Agree to use at least 1 highly effective form of contraception during study treatment and for at least 3 months after the last dose.

Exclusion Criteria:

* Any >Grade 1 persistent clinically significant toxicities from prior chemotherapy.
* Leukemic blast count >25 × 109/L. Hydroxyurea permitted to control leukocytosis.
* Known history of human immunodeficiency virus or active hepatitis B or active hepatitis C infection.
* Concomitant malignancies for which patients are receiving active therapy at the time of signing consent. Patients with adequately treated basal or squamous cell carcinoma of the skin, adequately treated carcinoma in situ (e.g., cervix), breast cancer receiving adjuvant endocrine therapy or prostate cancer not under active systemic treatment other than hormonal therapy may enroll irrespective of the time of diagnosis, with Medical Monitor approval.
* Known active central nervous system involvement by leukemia. Patients with previously diagnosed central nervous system leukemia are eligible if the central nervous system leukemia is under control and intrathecal treatment may continue throughout the study.
* Diagnosis of acute promyelocytic leukemia.
* Prior exposure to anticancer therapies including chemotherapy, radiotherapy or other investigational therapy, including targeted small molecule agents within 14 days of the first day of study treatment or within 5 half-lives prior to first dose of study treatment. Note that hydroxyurea up to 5 g daily × 3 days is permitted to reduce elevated white blood cell (WBC) count.
* Venetoclax exposure in more than 1 prior regimen.
* Prior exposure to biologic agents (e.g., monoclonal antibodies) for anti-neoplastic intent within 14 days prior to first dose of study drug.
* Prior hematopoietic stem cell transplantation.
* Malabsorption syndrome or other condition that precludes enteral route of administration.
* Pregnancy or lactation.
* Active uncontrolled systemic infection (viral, bacterial, or fungal).
* Ongoing treatment with strong or moderate CYP3A inhibitors or CYP3A inducers, P-gp inhibitors, or narrow therapeutic index P-gp substrates that cannot be discontinued at least 1 week prior to start of venetoclax dosing excluding antifungal prophylaxis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with dose-limiting toxicities assessed by CTCAE v5.0. | From the first day of treatment start until 30 days after treatment completion.
Number of patients with treatment-related adverse events assessed by CTCAE v5.0. | The first 28 days of study treatment (Cycle 1).
Recommended Phase 2 dose of DFP-10917 in combination with venetoclax (the dose at which <2 out of 6 patients experience a dose-limiting toxicity during the safety assessment period). | The first 28 days of study treatment (Cycle 1).

SECONDARY OUTCOMES:
The proportion of patients who achieve complete remission. | From the start of the study treatment to the first documented progression or death from any cause, whichever occurs first, assessed for up to 100 months.
The proportion of patients who achieve complete remission or complete remission with incomplete hematologic recovery. | From the start of the study treatment to the first documented progression or death from any cause, whichever occurs first, assessed for up to 100 months.
The proportion of patients achieving complete remission or complete remission with incomplete hematologic recovery, and morphologic leukemia-free state. | From the start of the study treatment to the first documented progression or death from any cause, whichever occurs first, assessed for up to 100 months.
Overall survival. | From the start of the study treatment to death from any cause, whichever occurs first, assessed for up to 100 months.
Progression-free survival. | From the start of the study treatment to the first documented progression or death from any cause, whichever occurs first, assessed for up to 100 months.
Maximum concentration of DFP-10917. | The first 15 days of study treatment.
Area under the curve of DFP-10917. | The first 15 days of study treatment.

OTHER OUTCOMES:
Volume of distribution of DFP-10917. | The first 15 days of study treatment.
Clearance of DFP-10917. | The first 15 days of study treatment.
Time to maximum concentration of venetoclax. | The first 15 days of study treatment.
Maximum concentration of venetoclax. | The first 15 days of study treatment.
Elimination half-life of venetoclax. | The first 15 days of study treatment.
Area under the curve of venetoclax. | The first 15 days of study treatment.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - UCI Chao Family Comprehensive Cancer Center, Orange, California
  - Atrium Health Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina
  - University of Vermont Cancer Center, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Undecided